CLINICAL TRIAL: NCT00801281
Title: First-line R-CVP vs R-CHOP Induction Immunochemotherapy for Indolent Lymphoma and R Maintenance.A Multicentre, Phase III Randomized Study by the PLRG.
Brief Title: First-line R-CVP vs R-CHOP Induction Immunochemotherapy for Indolent Lymphoma and R Maintenance.
Acronym: PLRG4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polish Lymphoma Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-CVP/CHOP
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma
Keywords: Lymphoma; Immunochemotherapy; Induction therapy; Maintenance therapy; Follicular lymphoma grade 1,2,3a; Marginal zone lymphoma, including MALT type; Small lymphocytic lymphoma (BM inv. <30%)
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-CVP (Active Comparator): Standard arm 1. R-CVP - Rituximab, Cyclophosphamide, Vincristine, Prednisone 2
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone 2
- R-CHOP (Experimental): Study arm 2. R-CHOP - Rituximab, Cyclophosphamide, Hydroxyldaunorubicine (doxorubicin), Oncovin (vincristine), Prednisone 1
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone 1

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 i.v. d. 1 q. 21 d.
  Other Names: MabThera
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 i.v. d. 1 q. 21 d.
  Other Names: Endoxan, Cytoxan
Drug: Doxorubicin — Doxorubicin 50 mg/m2 i.v. d. 1 q. 21 d.
  Other Names: Adriamycin
  Arms: R-CHOP
Drug: Vincristine — Vincristine 1.4 mg/m2 (max. 2 mg) i.v. d. 1 q. 21 d.
  Other Names: Oncovin
Drug: Prednisone 1 — Prednisone 100 mg p.o. d. 1-5 q. 21 d.
  Other Names: Deltasone
  Arms: R-CHOP
Drug: Prednisone 2 — Prednisone 40 mg/m2 p.o. d. 1-5 q. 21 d.
  Other Names: Deltasone
  Arms: R-CVP

SUMMARY:
Evaluation of event free survival (EFS) of patients treated with the study chemotherapy induction program: R-CHOP compared to the standard R-CVP regimen and response rates, time to best response, PFS, OS, neutropenic fever rate, infection rate, change in Ig levels, change in lymphocyte subpopulations counts in previously untreated indolent lymphoma patients in need of systemic treatment.

DETAILED DESCRIPTION:
Min. 3, max. 8 induction cycles. Maintenance with rituximab q. 2 months x 12/24 months, started 2 months after last chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed:
* Follicular lymphoma grade 1, 2, 3a
* Marginal zone lymphoma, including MALT type
* Small lymphocytic lymphoma (BM inv. < 30%)
* Lymphoplasmacytic lymphoma
* Clinical stage II-IV (Ann Arbor). Stage I is allowed if bulky (Ø > 7 cm) or if radiotherapy is not appropriate in judgment of treating physician
* Measurable lesion(s) in at least one site
* Patients previously untreated
* Patients presenting with symptoms requiring treatment:
* Progressive disease
* Symptoms related to tumor bulk
* Cytopenias related to bone marrow and/or spleen involvement B symptoms
* Age ≥ 18 years
* Performance status </=2
* Written informed consent

Exclusion Criteria:

* Grade 3b FL
* Transformed lymphoma
* CNS involvement
* Patient taking steroids for > 2 weeks during last 4 weeks at a dose equivalent to ≥ 20 mg prednisone
* Other malignancy
* Major surgery within 4 weeks
* Hb < 8 g/dl, ANC < 1.5 x 109/L, Plt <100 109/L unless due to lymphoma
* Impairment of renal function (creatinine > 1.5 x UNV) or liver function (total bilirubin 1.5 x UNV, SGOT > 2.5 x UNV not due to lymphoma
* Known infection, with HBV, HCV (acute < 6 mos. or chronic hepatitis) or HIV
* Serious underlying medical conditions
* Life expectancy < 6 months
* Known allergy to murine protein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-02; Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | +3 yrs

SECONDARY OUTCOMES:
Response Rate | +2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Walewski, Prof., Principal Investigator — Vice-president of PLRG; Maria Podolak-Dawidziak, Prof., Study Chair — PLRG Board Member; Beata Stella-Hołowiecka, Assoc. Prof., Study Chair — PLRG Member
Locations (12):
- Poland (12):
  - Podkarpacki Oncology Centre, Brzozów
  - Voivodeship Hospital, Oncology Ward, Elblag
  - Academic Clinical Centre, Hospital of Medical Academy, Clinic of Haematology and Transplantology, Gdansk
  - Silesian Medical University, Chair and Clinic of Haematology and Bone Marrow Transplantation, Katowice
  - Collegium Medicum Jagiellonian University, Clinic of Haematology, Krakow
  - Regional Oncology Centre, Ward of Proliferative Diseases, Lodz
  - Oncology Centre of Lublin Region, Lublin
  - Central Clinical Hospital, Ministry of Internal Matters and Administration; Clinic of Oncology, Haematology and Internal Diseases, Warsaw
  - Institute of Haematology and Transfusiology, Warsaw
  - M.Sklodowska-Curie Institute - Oncology Centre, Warsaw
  - Medical Academy in Wrocław; Chair and Clinic of Haematology, Blood Neoplasm and Bone Marrow Transplantation, Wroclaw
  - SP ZOZ Silesian Centre of Cellular Transplantation, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here to provide more information about this study: PLRG4 — http://www.plrg.coi.pl